CLINICAL TRIAL: NCT04811040
Title: A Phase 1b Randomized, Blinded, Proof-of-Concept Study to Evaluate the Safety and Efficacy of Broadly Neutralizing Antibodies (bNAbs) GS-5423 and GS-2872 in Combination With Capsid Inhibitor Lenacapavir (GS-6207) in Virologically Suppressed Adults With HIV-1 Infection
Brief Title: Study to Evaluate the Safety and Efficacy of Teropavimab and Zinlirvimab in Combination With Lenacapavir in Virologically Suppressed Adults With HIV-1 Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-536-5816
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — lenacapavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Clinical pharmacologist and sponsor are not masked to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Primary Cohort: Lenacapavir (LEN) + Teropavimab + Zinlirvimab 10 mg/kg (Experimental): Participants will receive a loading dose of 600 milligrams (mg) LEN orally on Day 1 and Day 2, along with 927 mg LEN as subcutaneous (SC) injection on Day 1. Thereafter, participants will receive 30 mg/kg teropavimab and then 10 mg/kg zinlirvimab as an intravenous (IV) infusion on Day 1.
  Interventions: Drug: Oral Lenacapavir; Drug: Subcutaneous Lenacapavir; Drug: Teropavimab; Drug: Zinlirvimab
- Primary Cohort: LEN + Teropavimab + Zinlirvimab 30 mg/kg (Experimental): Participants will receive a loading dose of 600 mg LEN orally on Day 1 and Day 2, along with 927 mg LEN as SC injection on Day 1. Thereafter, participants will receive 30 mg/kg teropavimab and then 30 mg/kg zinlirvimab as an IV infusion on Day 1.
  Interventions: Drug: Oral Lenacapavir; Drug: Subcutaneous Lenacapavir; Drug: Teropavimab; Drug: Zinlirvimab
- Pilot Cohort: LEN +Teropavimab +Zinlirvimab 10 mg/kg (Experimental): Participants will receive a loading dose of 600 mg LEN orally on Day 1 and Day 2, along with 927 mg LEN as SC injection on Day 1. Thereafter, participants will receive 30 mg/kg teropavimab and then 10 mg/kg zinlirvimab as an IV infusion on Day 1.
  Interventions: Drug: Oral Lenacapavir; Drug: Subcutaneous Lenacapavir; Drug: Teropavimab; Drug: Zinlirvimab
- Pilot Cohort: LEN +Teropavimab +Zinlirvimab 30 mg/kg (Experimental): Participants will receive a loading dose of 600 mg LEN orally on Day 1 and Day 2, along with 927 mg LEN as SC injection on Day 1. Thereafter, participants will receive 30 mg/kg teropavimab and then 30 mg/kg zinlirvimab as an IV infusion on Day 1.
  Interventions: Drug: Oral Lenacapavir; Drug: Subcutaneous Lenacapavir; Drug: Teropavimab; Drug: Zinlirvimab

INTERVENTIONS:
Drug: Oral Lenacapavir — Tablets administered without regard to food
  Other Names: GS-6207
Drug: Subcutaneous Lenacapavir — Administered in the abdomen via subcutaneous injections
  Other Names: GS-6207
Drug: Teropavimab — Administered intravenously
  Other Names: 3BNC117-LS; GS-5423
Drug: Zinlirvimab — Administered intravenously
  Other Names: 10-1074-LS; GS-2872

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of a combination of the broadly neutralizing antibodies (bNAbs) teropavimab (formerly GS-5423) and zinlirvimab (formerly GS-2872) in combination with the HIV capsid inhibitor lenacapavir (LEN).

ELIGIBILITY:
Key Inclusion Criteria:

* On first-line antiretroviral therapy (ART) for ≥ 2 years prior to screening. A change in ART regimen ≥ 28 days prior to screening for reasons other than virologic failure (VF) (eg, tolerability, simplification, drug-drug interaction profile) is allowed
* No documented historical resistance to the current ART regimen
* Plasma HIV-1 RNA < 50 copies/mL at screening
* Documented plasma HIV-1 RNA < 50 copies/mL for ≥ 18 months preceding the screening visit (or undetectable HIV-1 RNA level according to the local assay being used if the limit of detection is ≥ 50 copies/mL). Unconfirmed virologic elevations of ≥ 50 copies/mL (transient detectable viremia, or "blip") prior to screening are acceptable.
* Proviral phenotypic sensitivity to both teropavimab and zinlirvimab at screening by the PhenoSense mAb Assay (Monogram Biosciences) for inclusion in the Primary Cohort; sensitivity at screening by the PhenoSense mAb Assay (Monogram Biosciences) to 1 mAb, either teropavimab or zinlirvimab, within 18 months prior to enrollment for inclusion in the optional Pilot Cohort

  -- In both cohorts, teropavimab sensitivity is defined as 90% inhibitory concentration (IC90) ≤ 2 μg/mL; zinlirvimab sensitivity is defined as IC90 ≤ 2 μg/mL;
* Cluster determinant 4+ (CD4+) count nadir ≥ 350 cells/μL
* Screening CD4+ count ≥ 500 cells/μL
* Availability of a fully active alternative ART regimen, in the opinion of the investigator, in the event of discontinuation of the current ART regimen with development of resistance

Key Exclusion Criteria:

* Comorbid condition requiring ongoing immunosuppression
* Evidence of current hepatitis B virus (HBV) infection
* Evidence of current hepatitis C virus (HCV) infection (prior infection cleared spontaneously or with treatment is acceptable)
* History of opportunistic infection or illness indicative of Stage 3 HIV disease

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2023-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (23):
- United States (23):
  - Ruane Clinical Research Group Inc., Los Angeles, California
  - Mills Clinical Research, Los Angeles, California
  - One Community Health, Sacramento, California
  - UCSD AntViral Research Center (AVRC), San Diego, California
  - Yale University; School of Medicine; AIDS Program, New Haven, Connecticut
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - University of Miami Miller School of Medicine Schiff Center for Liver Disease, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Triple O Research Institute, P.A, West Palm Beach, Florida
  - Mercer University, Department of Internal Medicine, Macon, Georgia
  - Indiana CTSI Clinical Research Center, Indianapolis, Indiana
  - National Institutes of Health/Clinical Center, Bethesda, Maryland
  - Be Well Medical Center, Berkley, Michigan
  - AXCES Research Group, Santa Fe, New Mexico
  - Icahn School of Medicine at Mount Sinai-Clinical and Translational Research Center, New York, New York
  - NC TraCS Institute-CTRC; University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Brody School of Medicine at East Carolina University, ECU Adult Specialty Care, Greenville, North Carolina
  - Rosedale Health & Wellness, Huntersville, North Carolina
  - Perelman Center for Advanced Medicine at the Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - The Crofoot Research, INC., Houston, Texas
  - Peter Shalit, M.D., Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eron JJ, Cook PP, Mehrotra ML, Huang H, Caskey M, Crofoot GE, DeJesus E, Gorgos L, VanderVeen LA, Osiyemi OO, Brinson C, Collins SE. Lenacapavir Plus bNAbs for People with HIV and Susceptibility to Either Teropavimab or Zinlirvimab [Oral]. Conference on Retroviruses and Opportunistic Infections (CROI); 2024 3-6 March, Denver, CO.
- [Background] Eron JJ, Little SJ, Crofoot G, Cook P, Ruane PJ, Jayaweera D, VanderVeen LA, DeJesus E, Zheng Y, Mills A, Huang H, Waldman SE, Ramgopal M, Gorgos L, Collins SE, Baeten JM, Caskey M. Safety of teropavimab and zinlirvimab with lenacapavir once every 6 months for HIV treatment: a phase 1b, randomised, proof-of-concept study. Lancet HIV. 2024 Mar;11(3):e146-e155. doi: 10.1016/S2352-3018(23)00293-X. Epub 2024 Jan 30. PMID 38307098
- [Background] Eron J, Little SJ, Crofoot G, Cook P, Ruane PJ, Jayaweera D, DeJesus E, Walkman SE, Mehrotra ML, VanderVeen L, Huang H, Collins S, Baeten J, Caskey M. Lenacapavir with bNAbs Teropavimab (GS-5423) and Zinlirvimab (GS-2872) Dosed Every 6 Months in People with HIV [Oral 193]. Conference on Retroviruses and Opportunistic Infections (CROI); 2023 19-22 February, Seattle, WA
- [Background] Selzer L, VanderVeen LA, Parvangada A, Martin R, Collins SE, Mehrotra M, Callebaut C. Susceptibility Screening to bNAbs Teropavimab (GS-5423) and Zinlirvimab (GS-2872) in ART-Suppressed Participants [Poster]. Conference on Retroviruses and Opportunistic Infections (CROI); 2023 19-22 February; Seattle, WA
- [Background] Lisa Selzer, Sally Demirdjian, Ross Martin, Brie Falkard, Sean E. Collins, Joseph Eron, Laurie A. VanderVeen, Christian Callebaut. Resistance analyses during treatment of lenacapavir with broadly neutralizing antibodies in people with HIV (Poster WEPEB146) AIDS 2024; Munich, Germany
- [Background] Selzer L, VanderVeen LA, Parvangada A, Martin R, Collins SE, Mehrotra M, Callebaut C. Susceptibility Screening of HIV-1 Viruses to Broadly Neutralizing Antibodies, Teropavimab and Zinlirvimab, in People With HIV-1 Suppressed by Antiretroviral Therapy. J Acquir Immune Defic Syndr. 2025 Jan 1;98(1):64-71. doi: 10.1097/QAI.0000000000003528. PMID 39298557
- [Derived] Eron JJ, Cook PP, Mehrotra ML, Huang H, Caskey M, Crofoot GE, Gorgos L, VanderVeen LA, Zheng Y, Collins SE, Osiyemi OO, Brinson C, DeJesus E. Lenacapavir Plus 2 Broadly Neutralizing Antibodies, Teropavimab and Zinlirvimab, for People With HIV-1 Highly Susceptible to Either Teropavimab or Zinlirvimab. J Infect Dis. 2025 Jul 11;231(6):1440-1444. doi: 10.1093/infdis/jiaf159. PMID 40176256
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-536-5816

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States.
Pre-assignment Details: 124 participants were screened.
Groups:
- Primary Cohort: Lenacapavir (LEN)+Teropavimab+Zinlirvimab 10 mg/kg: Participants received a loading dose of 600 milligram (mg) LEN orally on Day 1 and Day 2, along with 927 mg LEN as subcutaneous (SC) injection on Day 1. Thereafter, participants received 30 milligram per kilogram (mg/kg) teropavimab and then 10 mg/kg zinlirvimab as an intravenous (IV) infusion on Day 1.
- Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg; Pilot Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg: Participants received a loading dose of 600 mg LEN orally on Day 1 and Day 2, along with 927 mg LEN as SC injection on Day 1. Thereafter, participants received 30 mg/kg teropavimab and then 30 mg/kg zinlirvimab as an IV infusion on Day 1.
- Pilot Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg: Participants received a loading dose of 600 mg LEN orally on Day 1 and Day 2, along with 927 mg LEN as SC injection on Day 1. Thereafter, participants received 30 mg/kg teropavimab and then 10 mg/kg zinlirvimab as an IV infusion on Day 1.
Period: Overall Study
Arm/Group | Primary Cohort: Lenacapavir (LEN)+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg | Pilot Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Pilot Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Started | 11 | 10 | 5 | 6
Completed | 8 | 9 | 5 | 6
Not Completed | 3 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Withdrew consent | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all randomized participants who have received at least one dose of study drug.
Groups:
- Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg; Pilot Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg: Participants received a loading dose of 600 mg LEN orally on Day 1 and Day 2, along with 927 mg LEN as SC injection on Day 1. Thereafter, participants received 30 mg/kg teropavimab and then 10 mg/kg zinlirvimab as an IV infusion on Day 1.
- Total: Total of all reporting groups
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg | Pilot Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Pilot Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg | Total
Number analyzed (Participants) | 11 | 10 | 5 | 6 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 5 | 6 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (9.8) | 41 (11.1) | 47 (15.1) | 46 (11.4) | 44 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 2 | 1 | 6
  Male | 11 | 7 | 3 | 5 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 2 | 1 | 10
  Not Hispanic or Latino | 7 | 7 | 3 | 5 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 7 | 5 | 3 | 3 | 18
  Race: Black or African American | 1 | 2 | 2 | 2 | 7
  Race: Other or More Than One Race | 1 | 2 | 0 | 1 | 4
  Race: Asian | 2 | 1 | 0 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 10 | 5 | 6 | 32

OUTCOME MEASURES:

1. Primary Outcome: Primary Cohort: Percentage of Participants Experiencing Treatment-Emergent Serious Adverse Events (SAEs)
Description: A treatment emergent SAE was defined as an event that, at any dose, resulted in the following: death; life-threatening situation; in-patient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; a congenital anomaly/birth defect; a medically important event or reaction: such events may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes constituting SAEs. These events had an onset date on or after the study drug start date and prior to the last exposure date of long-acting (LA) regimen period for the LA regimen period analysis. The long acting regimen period included participants who were randomized and received at least one dose of the complete LA study drug regimen (ie, SC LEN + Teropavimab + Zinlirvimab).
Time Frame: Day 1 up to Week 26
Population: The Safety Analysis Set for the LA regimen included all randomized participants who had received at least 1 dose of the complete LA study drug regimen (ie, SC LEN + Teropavimab + Zinlirvimab).
Measure: Number; unit: percentage of participants
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 10 | 10
percentage of participants | 0 | 0

2. Secondary Outcome: Primary Cohort: Percentage of Participants With Human Immunodeficiency Virus- 1 Ribonucleic Acid (HIV-1 RNA) < 50 Copies/mL at Week 26 as Determined by the US Food and Drug Administration (FDA)-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 26 was analyzed using the snapshot algorithm, which defined a participant's virologic outcome and included participants who had the last available on-treatment HIV-1 RNA < 50 copies/mL in the Week 26 analysis window. Week 26 window was between Days 176 and 224 (inclusive).
Time Frame: Week 26
Population: The Full Analysis Set included all randomized participants who had received at least 1 dose of the complete LA study drug regimen (ie, SC LEN + Teropavimab + Zinlirvimab) without major protocol violation (defined as meeting exclusion criterion of having chronic hepatitis B virus infection).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 10 | 10
percentage of participants | 90.0 [55.5 to 99.7] | 90.0 [55.5 to 99.7]

3. Secondary Outcome: Primary Cohort: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 26 as Determined by the US FDA-defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 26 was analyzed using the snapshot algorithm, which defined a participant's virologic outcome and included participants a) who had the last available on-treatment HIV-1 RNA ≥ 50 copies/mL in the Week 26 analysis window; b) who did not have on-treatment HIV-1 RNA data in the Week 26 analysis window and i) discontinued study drug prior to or in the Week 26 analysis window due to lack of efficacy, or ii) discontinued study drug prior to or in the Week 26 analysis window due to AE or death and had the last available on-treatment HIV-1 RNA ≥ 50 copies/mL, or iii) discontinued study drug prior to or in the Week 26 analysis window due to reasons other than AE, death, or lack of efficacy and had the last available on-treatment HIV-1 RNA ≥ 50 copies/mL.
  Week 26 window was between Days 176 and 224 (inclusive).
Time Frame: Week 26
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 10 | 10
percentage of participants | 10.0 [0.3 to 44.5] | 0 [0.0 to 30.8]

4. Secondary Outcome: Primary Cohort: Percentage of Participants With Positive Anti-Teropavimab Antibodies
Description: Anti-teropavimab antibodies positive participants are participants with positive treatment-emergent anti-drug antibody.
Time Frame: Week 26
Population: Anti-teropavimab Immunogenicity Analysis Set included all randomized participants who had received at least 1 dose of study drug and have had at least 1 nonmissing value for anti-teropavimab evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 10 | 10
percentage of participants | 50.0 | 10.0

5. Secondary Outcome: Primary Cohort: Percentage of Participants With Positive Anti-zinlirvimab Antibodies
Description: Anti-zinlirvimab antibodies positive participants are participants with positive treatment-emergent anti-drug antibody.
Time Frame: Week 26
Population: Anti-zinlirvimab Immunogenicity Analysis Set included all randomized participants who had received at least 1 dose of study drug and have had at least 1 nonmissing value for anti- zinlirvimab evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 10 | 10
percentage of participants | 40.0 | 20.0

6. Secondary Outcome: Primary Cohort: Change From Baseline in Cluster Determinant 4+ (CD4+) Cell Count at Week 26
Time Frame: Baseline; Week 26
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells per microliter (cells/µL)
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 10 | 10
cells per microliter (cells/µL)
  Baseline | 903 (303.7) | 1086 (333.6)
  Week 26: number analyzed (Participants) | 8 | 9
  Week 26 | -25 (241.6) | -5 (162.2)

7. Secondary Outcome: Primary Cohort: Number of Participants Who Develop Treatment-Emergent Resistance to LEN, Teropavimab, and Zinlirvimab
Description: Participants in the Resistance Analysis Population analyzed for this outcome included any participant who had received 1 dose of study drug, maintained their study drug regimen, and met one of the following virologic failure criteria:
  * Participants with HIV-1 RNA >/= 200 copies/mL on 2 consecutive visits
  * Participants with HIV-1 RNA >/= 200 copies/mL at study discontinuation or Week 26.
Time Frame: Day 1 up to Week 26
Population: Participants in the Resistance Analysis Population included those who experienced virologic failure through Week 26.
Measure: Count of Participants; unit: Participants
Groups:
- Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg: Participants received a loading dose of 600 mg LEN orally on Day 1 and Day 2, along with 927 mg LEN as SC injection on Day 1. Thereafter, participants were administered 30 mg/kg teropavimab and then 10 mg/kg zinlirvimab intravenously on Day 1.
- Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg: Participants received a loading dose of 600 mg LEN orally on Day 1 and Day 2, along with 927 mg LEN as SC injection on Day 1. Thereafter, participants were administered 30 mg/kg teropavimab and then 30 mg/kg zinlirvimab intravenously on Day 1.
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 1 | 0
Participants
  Participants who developed resistance to LEN | 1 |
  Participants who developed resistance to Teropavimab | 0 |
  Participants who developed resistance to Zinlirvimab | 0 |

8. Secondary Outcome: Primary Cohort: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were those adverse events that began on or after the first dose date of study drug and prior to last exposure date of LA regimen from participants who prematurely discontinued study or completed study, or any adverse events led to premature study drug discontinuation.
Time Frame: Day 1 up to Week 26
Population: Participants in the Safety Analysis Set for the LA regimen were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 10 | 10
percentage of participants | 90 | 100

9. Secondary Outcome: Primary Cohort: Pharmacokinetic (PK) Parameter: AUC0-26 of Teropavimab
Description: AUC0-26 is defined as the concentration of drug over time from Week zero to Week 26.
Time Frame: Predose and at End of Infusion (EOI) of teropavimab and zinlirvimab on Day 1; Weeks 4, 8, 12, 16, 20, 24, 26
Population: The Teropavimab PK Analysis Set included all randomized participants who had received at least 1 dose of study drug, and had at least 1 nonmissing teropavimab concentration value reported by the PK laboratory test.
Measure: Mean (Standard Deviation); unit: day* μg/mL
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 10 | 10
day* μg/mL | 30500 (2270) | 31600 (3750)

10. Secondary Outcome: Primary Cohort: PK Parameter: AUC0-26 of Zinlirvimab
Description: AUC0-26 is defined as the concentration of drug over time from Week zero to Week 26.
Time Frame: Predose and at EOI of teropavimab and zinlirvimab on Day 1; Weeks 4, 8, 12, 16, 20, 24, 26
Population: The Zinlirvimab PK Analysis Set included all randomized participants who had received at least 1 dose of study drug, and had at least 1 nonmissing zinlirvimab concentration value reported by the PK laboratory test. Participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: day* μg/mL
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 9 | 9
day* μg/mL | 14800 (2090) | 46100 (4180)

11. Secondary Outcome: Primary Cohort: PK Parameter: AUClast of Teropavimab
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Time Frame: Predose and at EOI of teropavimab and zinlirvimab on Day 1; Weeks 4, 8, 12, 16, 20, 24, 26, 38, 52, up to end of study (up to Week 55)
Population: Participants in the Teropavimab PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: day* μg/mL
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 10 | 10
day* μg/mL | 32900 (3140) | 34400 (5500)

12. Secondary Outcome: Primary Cohort: PK Parameter: AUClast of Zinlirvimab
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Time Frame: as for outcome 11
Population: Participants in the Zinlirvimab PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: day* μg/mL
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 9 | 9
day* μg/mL | 17100 (2640) | 54700 (5290)

13. Secondary Outcome: Primary Cohort: PK Parameter: T1/2 of LEN
Description: T1/2 is defined as the estimate of the terminal elimination half-life of the drug.
Time Frame: as for outcome 11
Population: The LEN PK Analysis Set included all randomized participants who had received at least 1 dose of study drug, and had at least 1 nonmissing LEN concentration value reported by the PK laboratory test. Participants with available data were analyzed.
Measure: Median (Full Range); unit: day
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 8 | 9
day | 65.8 [33.9 to 99.3] | 69.8 [55.1 to 140]

14. Secondary Outcome: Primary Cohort: PK Parameter: T1/2 of Teropavimab
Description: T1/2 is defined as the estimate of the terminal elimination half-life of the drug.
Time Frame: as for outcome 11
Population: Participants in the Teropavimab PK Analysis Set were analyzed.
Measure: Median (Full Range); unit: day
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 10 | 10
day | 65.2 [54.3 to 78.3] | 70.5 [57.5 to 89.6]

15. Secondary Outcome: Primary Cohort: PK Parameter: T1/2 of Zinlirvimab
Description: T1/2 is defined as the estimate of the terminal elimination half-life of the drug.
Time Frame: as for outcome 11
Population: Participants in the Zinlirvimab PK Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: day
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 10 | 9
day | 76.7 [43.4 to 113] | 84.5 [71.6 to 149]

16. Secondary Outcome: Primary Cohort: PK Parameter: Cmax of Teropavimab
Description: Cmax is defined as the maximum observed concentration of drug.
Time Frame: as for outcome 11
Population: Participants in the Teropavimab PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 10 | 10
μg/mL | 1090 (160) | 1090 (222)

17. Secondary Outcome: Primary Cohort: PK Parameter: Cmax of Zinlirvimab
Description: Cmax is defined as the maximum observed concentration of drug.
Time Frame: as for outcome 11
Population: Participants in the Zinlirvimab PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 9 | 9
μg/mL | 378 (57.5) | 1110 (187)

18. Secondary Outcome: Primary Cohort: PK Parameter: Tmax of Teropavimab
Description: Tmax is defined as the time (observed time point) of Cmax.
Time Frame: as for outcome 11
Population: Participants in the Teropavimab PK Analysis Set were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 10 | 10
hours | 1.16 [1.02 to 2.75] | 2.24 [0.983 to 2.83]

19. Secondary Outcome: Primary Cohort: PK Parameter: Tmax of Zinlirvimab
Description: Tmax is defined as the time (observed time point) of Cmax.
Time Frame: as for outcome 11
Population: Participants in the Zinlirvimab PK Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 9 | 9
hours | 1.10 [0.983 to 1.37] | 1.00 [0.850 to 1.23]

20. Secondary Outcome: Primary Cohort: PK Parameter: Tlast of LEN
Description: Tlast is defined as the time (observed time point) of Clast (the last observable concentration of drug).
Time Frame: as for outcome 11
Population: Participants in the LEN PK Analysis Set were analyzed.
Measure: Median (Full Range); unit: day
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 10 | 10
day | 364 [168 to 366] | 364 [84.0 to 373]

21. Secondary Outcome: Primary Cohort: PK Parameter: Tlast of Teropavimab
Description: Tlast is defined as the time (observed time point) of Clast (the last observable concentration of drug).
Time Frame: as for outcome 11
Population: Participants in the Teropavimab PK Analysis Set were analyzed.
Measure: Median (Full Range); unit: day
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 10 | 10
day | 364 [168 to 366] | 364 [83.9 to 373]

22. Secondary Outcome: Primary Cohort: PK Parameter: Tlast of Zinlirvimab
Description: Tlast is defined as the time (observed time point) of Clast (the last observable concentration of drug).
Time Frame: as for outcome 11
Population: Participants in the Zinlirvimab PK Analysis Set were analyzed.
Measure: Median (Full Range); unit: day
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 10 | 10
day | 364 [168 to 366] | 364 [83.9 to 373]

23. Secondary Outcome: Primary Cohort: PK Parameter: C26week of LEN
Description: C26week is the concentration at week 26.
Time Frame: Week 26
Population: Participants in the LEN PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 8 | 8
ng/mL | 27.2 (17.4) | 22.5 (17.0)

24. Secondary Outcome: Primary Cohort: PK Parameter: C26week of Teropavimab
Description: C26week is the concentration at week 26.
Time Frame: Week 26
Population: Participants in the Teropavimab PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 8 | 8
μg/mL | 38.4 (5.89) | 42.7 (6.49)

25. Secondary Outcome: Primary Cohort: PK Parameter: C26week of Zinlirvimab
Description: C26week is the concentration at week 26.
Time Frame: Week 26
Population: Participants in the Zinlirvimab PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
Number analyzed (Participants) | 8 | 8
μg/mL | 27.2 (6.44) | 84.6 (27.1)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Up to 55.9 weeks; Adverse Events: Up to 51.1 weeks
Description: All-cause Mortality: All Randomized Analysis Set included all participants who were randomized into the study.
  Adverse Event: The Safety Analysis Set included all randomized participants who had received at least one dose of study drug.
Arm/Group | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg | Pilot Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg | Pilot Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/11 | 0/10 | 1/5 | 0/6
Other Adverse Events (participants affected / at risk) | 9/11 | 10/10 | 4/5 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg (N=11) | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg (N=10) | Pilot Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg (N=5) | Pilot Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg (N=6)
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg (N=11) | Primary Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg (N=10) | Pilot Cohort: LEN+Teropavimab+Zinlirvimab 10 mg/kg (N=5) | Pilot Cohort: LEN+Teropavimab+Zinlirvimab 30 mg/kg (N=6)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Glossitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 1 | 0 | 0
Injection site discolouration (General disorders) | 1 | 1 | 0 | 0
Injection site erythema (General disorders) | 4 | 3 | 0 | 2
Injection site induration (General disorders) | 2 | 4 | 0 | 3
Injection site inflammation (General disorders) | 0 | 1 | 0 | 0
Injection site mass (General disorders) | 3 | 1 | 0 | 0
Injection site nodule (General disorders) | 4 | 2 | 1 | 1
Injection site oedema (General disorders) | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 5 | 5 | 0 | 2
Injection site paraesthesia (General disorders) | 1 | 0 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 2
Injection site reaction (General disorders) | 1 | 1 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0
Bacterial vulvovaginitis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 4 | 1 | 1 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 1 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0
Gonorrhoea (Infections and infestations) | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0
Injection site cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Oropharyngeal gonococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngeal chlamydia infection (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Secondary syphilis (Infections and infestations) | 0 | 0 | 1 | 0
Shigella infection (Infections and infestations) | 1 | 0 | 0 | 0
Syphilis (Infections and infestations) | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 0 | 1
Varicella zoster virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myokymia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Bladder discomfort (Renal and urinary disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Genital lesion (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT04811040/Prot_000.pdf
  • Statistical Analysis Plan: Week 26 Analysis (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT04811040/SAP_001.pdf
  • Statistical Analysis Plan: Final Analysis (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT04811040/SAP_002.pdf